CLINICAL TRIAL: NCT02126852
Title: Comparison of AMG (Acceleromyography) and EMG (Electromyography) to Avoid Postoperative Residual Paralysis After General Anesthesia
Brief Title: Comparison of AMG and EMG to Avoid Residual Paralysis After General Anesthesia
Acronym: CAMEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAMEM
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Observation of Neuromuscular Block; Respiratory Paralysis; Anaesthesia
Keywords: residual paralysis,neuromuscular blockade,acceleromyography,electromyography
MeSH Terms: conditions — Respiratory Paralysis | interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG (one-dimensionally) versus EMG (Experimental): Neuromuscular monitoring in patients scheduled for surgery under general anesthesia
  Interventions: Device: Acceleromyography (AMG, one-dimensionally); Device: Electromyography (EMG)
- AMG (three-dimensionally) versus EMG (Experimental): Neuromuscular monitoring in patients scheduled for surgery under general anesthesia
  Interventions: Device: Acceleromyography (AMG, three-dimensionally); Device: Electromyography (EMG)

INTERVENTIONS:
Device: Acceleromyography (AMG, one-dimensionally) — Neuromuscular monitoring
  Arms: AMG (one-dimensionally) versus EMG
Device: Acceleromyography (AMG, three-dimensionally) — Neuromuscular monitoring
  Arms: AMG (three-dimensionally) versus EMG
Device: Electromyography (EMG) — Neuromuscular monitoring

SUMMARY:
This study evaluates three different neuromuscular monitoring devices (acceleromyography, one- or three-dimensional, and electromyography) with regard to their precision to detect residual paralysis after injection of neuromuscular blocking agents and recurrence of paralysis after administration of reversal agents in a clinical setting.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are routinely used as standard part of a modern, balanced anesthesia regime. A residual duration of action exceeding the end of surgery, also called residual neuromuscular paralysis, is a common undesired side effect and increases the risk for postoperative pulmonary complications such as aspiration or pneumonia delaying patients' discharge from the post-anesthesia care unit. To limit the incidence of residual paralysis in daily anesthesia care, quantitative neuromuscular monitoring is recommended after injection of NMBAs. If a residual effect of a NMBA is detected at the end of surgery, reversal agents such as cholinesterase inhibitors, e.g. neostigmine or a selective relaxant binding agent, e.g. sugammadex can be administered. However, if reversal agents are not adequately dosed, the risk for a residual neuromuscular blockade re-occurs. Accordingly, neuromuscular monitoring is also useful to control the action of the administered reversal agents.

Although several techniques of neuromuscular monitoring are established in clinical practice, electromyography (EMG) and acceleromyography (AMG) are the most common quantitative neuromuscular monitoring devices. Electromyography, the gold standard for detecting residual neuromuscular block, is based on measuring summarized spikes of evoked muscle contractions. Acceleromyography measuring the acceleration of evoked muscle contraction is also commercially available and easy to use. This acceleration, however, can be measured both one-dimensionally and three-dimensionally.

This study evaluates the three described neuromuscular monitoring devices with regard to their precision to detect residual paralysis after administration of NMBAs and recurrence of neuromuscular blockade after administration of reversal agents in a clinical setting. We plan to include and randomize a total of 200 patients. The study participants will be recruited from patients scheduled for surgery at the Klinikum rechts der Isar der Technischen Universität München, Munich, Germany. In each patient, acceleromyography (either one- or three-dimensional) will be compared with the calibrated electromyography. The findings will help to indicate which neuromuscular monitoring device is most suitable for detecting residual paralysis and recurrent neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA physical status I-III
* Patients older than 18 years
* General anesthesia with the use of the neuromuscular blocking agent rocuronium
* Expected duration of surgery more than 2 hours
* Patients having given informed consent to the study

Exclusion Criteria:

* Known or suspected allergy towards anesthetics/sugammadex or rocuronium
* Pregnant and breastfeeding women
* Known or suspected neuromuscular disease (Multiple sclerosis, myasthenia gravis)
* Anatomic and functional malformations with expected difficult intubation
* body mass index >35kg/m2
* Contraindication for the use of rocuronium or sugammadex
* Malignant hyperthermia
* Patients with a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
This study evaluates the precision and agreement of TOF-ratios obtained with acceleromyography and electromyography during residual neuromuscular paralysis | during surgery (2 hours)

SECONDARY OUTCOMES:
Incidence of re-occurrence of neuromuscular block after administration of reversal agents measured with acceleromyography and electromyography | during surgery (2 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, M.D., Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München, Germany
Locations (2):
- Germany (2):
  - Department of Anesthesiology, Munich
  - Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duvaldestin P, Kuizenga K, Saldien V, Claudius C, Servin F, Klein J, Debaene B, Heeringa M. A randomized, dose-response study of sugammadex given for the reversal of deep rocuronium- or vecuronium-induced neuromuscular blockade under sevoflurane anesthesia. Anesth Analg. 2010 Jan 1;110(1):74-82. doi: 10.1213/ANE.0b013e3181c3be3c. Epub 2009 Nov 21. PMID 19933538
- [Background] Liang SS, Stewart PA, Phillips S. An ipsilateral comparison of acceleromyography and electromyography during recovery from nondepolarizing neuromuscular block under general anesthesia in humans. Anesth Analg. 2013 Aug;117(2):373-9. doi: 10.1213/ANE.0b013e3182937fc4. Epub 2013 Jul 2. PMID 23821356
- [Background] Eleveld DJ, Kuizenga K, Proost JH, Wierda JM. A temporary decrease in twitch response during reversal of rocuronium-induced muscle relaxation with a small dose of sugammadex. Anesth Analg. 2007 Mar;104(3):582-4. doi: 10.1213/01.ane.0000250617.79166.7f. PMID 17312212
- [Background] Puhringer FK, Gordon M, Demeyer I, Sparr HJ, Ingimarsson J, Klarin B, van Duijnhoven W, Heeringa M. Sugammadex rapidly reverses moderate rocuronium- or vecuronium-induced neuromuscular block during sevoflurane anaesthesia: a dose-response relationship. Br J Anaesth. 2010 Nov;105(5):610-9. doi: 10.1093/bja/aeq226. Epub 2010 Sep 28. PMID 20876699